CLINICAL TRIAL: NCT03723759
Title: A Trial Investigating the Pharmacokinetic Properties of Five Formulations of Fast-acting Insulin Aspart 200 U/mL in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Research Study Looking at How Faster Aspart Injected in Double Concentration Works in the Body of People With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1200-4431; U1111-1209-2099 (Other: World Health Organization (WHO)); 2018-000593-30 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is asked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group A (Experimental): Participants will be allocated to a treatment sequence consisting of 5 formulations of faster aspart 200 U/mL and faster aspart 100 U/mL in following sequence:
  formulation D, faster aspart 100 U/mL, formulation B, formulation A, formulation C, formulation E.
  The dosing visits will be separated by wash-out periods (2-21 days).
  Interventions: Drug: Faster Aspart 200 U/mL; Drug: Faster aspart 100 U/mL
- Group B (Experimental): Participants will be allocated to a treatment sequence consisting of 5 formulations of faster aspart 200 U/mL and faster aspart 100 U/mL in following sequence:
  formulation C, formulation B, formulation D, formulation E, formulation A, faster aspart 100 U/mL.
  The dosing visits will be separated by wash-out periods (2-21 days).
  Interventions: Drug: Faster Aspart 200 U/mL; Drug: Faster aspart 100 U/mL
- Group C (Experimental): Participants will be allocated to a treatment sequence consisting of 5 formulations of faster aspart 200 U/mL and faster aspart 100 U/mL in following sequence:
  formulation E, formulation C, formulation A, formulation B, faster aspart 100 U/mL, formulation D.
  The dosing visits will be separated by wash-out periods (2-21 days).
  Interventions: Drug: Faster Aspart 200 U/mL; Drug: Faster aspart 100 U/mL
- Group D (Experimental): Participants will be allocated to a treatment sequence consisting of 5 formulations of faster aspart 200 U/mL and faster aspart 100 U/mL in following sequence:
  formulation A, formulation D, formulation C, faster aspart 100 U/mL, formulation E, formulation B.
  The dosing visits will be separated by wash-out periods (2-21 days).
  Interventions: Drug: Faster Aspart 200 U/mL; Drug: Faster aspart 100 U/mL
- Group E (Experimental): Participants will be allocated to a treatment sequence consisting of 5 formulations of faster aspart 200 U/mL and faster aspart 100 U/mL in following sequence:
  faster aspart 100 U/mL, formulation A, formulation E, formulation D, formulation B, formulation C.
  The dosing visits will be separated by wash-out periods (2-21 days).
  Interventions: Drug: Faster Aspart 200 U/mL; Drug: Faster aspart 100 U/mL
- Group F (Experimental): Participants will be allocated to a treatment sequence consisting of 5 formulations of faster aspart 200 U/mL and faster aspart 100 U/mL in following sequence:
  formulation B, formulation E, faster aspart 100 U/mL, formulation C, formulation D, formulation A.
  The dosing visits will be separated by wash-out periods (2-21 days).
  Interventions: Drug: Faster Aspart 200 U/mL; Drug: Faster aspart 100 U/mL

INTERVENTIONS:
Drug: Faster Aspart 200 U/mL — A single dose (0.15 U/kg) of five formulations of fast-acting insulin aspart 200 U/mL (formulations A, B, C, D, E) in a sequential manner via subcutaneous injection.
Drug: Faster aspart 100 U/mL — A single dose (0.15 U/kg) of fast-acting insulin aspart 100 U/mL via subcutaneous injection.

SUMMARY:
This study is looking at how five different formulations of faster aspart 200 U/mL reach and stay in the blood after injection. The purpose is to find a formulation that behaves similarly to the reference product called faster aspart 100 U/mL (marketed as Fiasp®). The participant will get all five formulations and the reference product. The order in which the participant gets them is decided by chance. The participant will get each medicine once during the study meaning that the participant will get a total of six injections with study medicine. The medicine will be injected under the skin in the stomach. The study will last for about 2 to 21 weeks depending on individual visit schedule. The participant will have nine clinic visits with the study doctor (including the one in which the participant give consent).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at the time of signing informed consent
* Diagnosed with type 1 diabetes mellitus greater than or equal to 1 year prior to the day of screening
* Treated with multiple daily insulin injections or continuous subcutaneous insulin infusion greater than or equal to 1 year prior to the day of screening

Exclusion Criteria:

* Participation in any clinical trial of an approved or non-approved investigational medicinal product within 90 days before screening in this trial
* Blood donation, plasma donation or blood draw, defined as any of the below: In excess of 400 mL within the past 90 days prior to the day of screening OR In excess of 50 mL within the past 30 days prior to the day of screening
* Use of tobacco and nicotine products, defined as any of the below: Smoking more than 1 cigarette or the equivalent per day OR Not able or willing to refrain from smoking and use of nicotine substitute products during the in-house periods

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2018-10-26 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
AUCIAsp,0h-t - Area under the serum insulin aspart concentration-time curve from 0 to t hours after investigational medicinal product (IMP) administration, where t is end of exposure | 0 to 10 hours after IMP administration
  Measured in pmol*h/L

SECONDARY OUTCOMES:
AUCIAsp,0-1h - Area under the serum insulin aspart concentration-time curve from 0 to 1 hour after IMP administration | 0 to 1 hour after IMP administration
  Measured in pmol*h/L
AUCIAsp,0-2h - Area under the serum insulin aspart concentration-time curve from 0 to 2 hours after IMP administration | 0 to 2 hours after IMP administration
  Measured in pmol*h/L
AUCIAsp,0-inf - Area under the serum insulin aspart concentration-time curve from 0 hours after IMP administration to infinity | 0 to 10 hours after IMP administration
  Measured in pmol*h/L
Cmax,IAsp - Maximum observed serum insulin aspart concentration | 0 to 10 hours after IMP administration
  Measured in pmol/L
tmax,IAsp - Time to maximum observed serum insulin aspart concentration | 0 to 10 hours after IMP administration
  Measured in minutes
Number of adverse events in the treatment emergent period | 0 to 2 days after IMP administration
  Count of events
Number of local reactions at the injection site in the treatment emergent period | 0 to 2 days after IMP administration
  Count of injection site reactions
Number of hypoglycaemic episodes in the treatment emergent period | 0 to 16 hours after IMP administration
  Count of hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com